CLINICAL TRIAL: NCT04418778
Title: The Building Empowerment and Resilience Therapeutic Program for Women With a History of Trauma
Brief Title: The BEAR Therapeutic Program for Women
Status: Active, not recruiting | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jennifer Keller, Clinical Professor, Stanford University
Other Study IDs: 54562
Record Dates: First submitted 2020-05-29; First posted 2020-06-05 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Trauma, Psychological; Depression, Anxiety; PTSD
Keywords: empowerment; therapeutic intervention
MeSH Terms: conditions — Psychological Trauma; Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic; Empowerment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BEAR intervention group: BEAR Therapeutic group for women who have experienced interpersonal trauma
  Interventions: Behavioral: BEAR
- Control Condition: Treatment as usual group, women participating in individual or group therapy but not taking the BEAR group

INTERVENTIONS:
Behavioral: BEAR — Building Empowerment and Resilience Therapy group
  Groups: BEAR intervention group

SUMMARY:
The current study aims to test a novel therapeutic intervention for women who have a history of interpersonal trauma. The Building Empowerment and Resilience (BEAR) Therapeutic group incorporates psychological skills, psychoeducation, and physical empowerment training, all within a therapeutic process. It will be implemented iwith women who have experienced interpersonal trauma (physical, sexual, or emotional abuse/neglect). The investigators aim to understand how this program effects one's self-efficacy and whether the program can reduce rates mental health problems (such as depression and anxiety) and reduce the rates of revictimization. Women who participate in the BEAR group must be able to attend in-person sessions. The control group can be remote.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages 18-70
2. History of physical, sexual, and/or emotional abuse/neglect/violence, with subsequent interpersonal or psychological distress (e.g., depression or anxiety) related to this history.

Exclusion Criteria:

1. Active, significant substance abuse
2. Significant medical conditions that would preclude safe participation in the study
3. High levels of depression with significant suicide risk
4. Psychiatric instability
5. History of assaultive behavior or is judged to be at potential risk to assault others.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female identified participants
Study Population: Women who have experienced interpersonal violence broadly defined
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in Coping Self-Efficacy Scale (CSES) | baseline to post-group (3 months)
  The CSES is designed to measure an individual's perception of her competence to carry out coping strategies effectively when faced with a challenge or threat.
Trauma Symptom Inventory-II (TSI-2). | baseline to post-group (3 months)
  The TSI-2 is a self-report measure of trauma-related symptoms and behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States